CLINICAL TRIAL: NCT05379829
Title: Pharmacokinetics, Pharmacodynamics and Safety of Ziltivekimab Versus Placebo in Chinese Participants With Chronic Kidney Disease and Systemic Inflammation
Brief Title: A Research Study of How the Medicine Ziltivekimab Works in the Body of Chinese Men and Women With Kidney Disease and Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6018-4889; U1111-1266-5585 (Other: WHO)
Record Dates: First submitted 2022-05-15; First posted 2022-05-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease and Systemic Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ziltivekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ziltivekimab 15 mg (Experimental): Participants will receive ziltivekimab at weeks 0, 4 and 8.
  Interventions: Drug: Ziltivekimab
- Placebo (Placebo Comparator): Participants will receive placebo at weeks 0, 4 and 8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziltivekimab — Participants will be administered 3 doses subcutaneously (s.c.) every four weeks (Q4W).
  Arms: Ziltivekimab 15 mg
Drug: Placebo — Participants will be administered 3 doses s.c. Q4W.
  Arms: Placebo

SUMMARY:
This study is conducted to see how the ziltivekimab works in the body of Chinese people with chronic kidney disease and systemic inflammation. Participants will either get ziltivekimab (active medicine) or placebo (a dummy medicine which has no effect on the body. Participants' chance of getting ziltivekimab or placebo is the same.

Participants will get their study medicine in a pre-filled syringe. The study doctor or staff will do 3 injections of study medicine during clinical visits.

The study is expected to last for about 6 months. Participants will have blood and urine samples taken at all of the clinic visits. Participants will have their heart examined using electrodes (electrocardiogram).

Women cannot take part if pregnant, breast-feeding or planning to get pregnant during the study period.

ELIGIBILITY:
Inclusion criteria:

1. Estimated glomerular filtration rate (eGFR) greater than or equal 15 and less than 60 mL/min/1.73 m^2 [Millilitre/minute] (using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation)
2. Serum high-sensitivity C-reactive protein (hs-CRP) greater than or equal to 2 mg/L [Milligram Per Litre] at screening (visit 1).

Exclusion criteria:

Laboratory values

1. Absolute neutrophil count less than 2×10^9/Litre at screening (visit 1).
2. Platelet count less than 120×10^9/Litre at screening (visit 1).
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 × upper limit of normal at screening (visit 1).

Medical conditions

1. Clinical evidence of, or suspicion of, active infection at the discretion of the investigator.
2. History of gastrointestinal perforation. (Note: History of perforated appendicitis more than 5 years prior to screening (visit 1) is not exclusionary).
3. History of active diverticulitis in the 5 years prior to randomization (visit 2).
4. History of inflammatory bowel disease that has been clinically active during the 12 months prior to randomization (visit 2).
5. Myocardial infarction, stroke, hospitalization for unstable angina pectoris, or transient ischemic attack within 60 days prior to randomization (visit 2).
6. Planned coronary, carotid or peripheral artery revascularization known on the day of screening (visit 1).
7. Major cardiac surgical, non-cardiac surgical, or major endoscopic procedure (thoracoscopic or laparoscopic) within the past 60 days prior to randomization (visit 2) or any major surgical procedure planned at the time of randomization (visit 2). Prior or current medication

1. Use of preventive systemic antibiotics, systemic antivirals, or systemic antifungals at screening (visit 1). (Note: "Systemic" is defined as oral or intravenous (i.v.) administered drugs that are absorbed into the circulation).

2. Use of systemic immunosuppressive drugs (both small molecules and biologics) or biologic disease modifying anti-rheumatic drugs (DMARDs including both biologic DMARDs like anti-TNF-alpha and conventional DMARDs like methotrexate) at screening (visit 1) or anticipated chronic use of such drugs any time during the study. (Note: Use of otic, ophthalmic, inhaled, and topical corticosteroids or local corticosteroid injections are not exclusionary).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Area under the ziltivekimab plasma concentration-time curve in a 4-week dosing interval, multiple doses [MD] (AUCτ,MD) | During 3rd dosing interval (week 8 to week 12)
  Nanograms per millilitre*days (ng/mL*days)

SECONDARY OUTCOMES:
Change in hs-CRP (high-sensitivity C-reactive protein | From baseline (week 0) to end of treatment (week 12)
  Milligrams per millilitre (mg/L)
Area under the ziltivekimab plasma concentration-time curve in a 4-week dosing interval, single dose [SD] | During 1st dosing interval (day 0 to week 4)
  ng/mL*days
Maximum plasma concentration of ziltivekimab after 3rd dose (Cmax,MD) | After last dose (week 8) to end of study (week 20)
  ng/mL
Elimination half-life (t½) | After last dose (week 8) to end of study (week 20)
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (7):
- China (7):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinses People's Liberation Army General Hospital-Nephrology, Beijing, Beijing Municipality
  - Zhongda Hospital Southeast University-Nephrology, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University-Neurology, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University-Endocrinology, Suzhou, Jiangsu
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com